CLINICAL TRIAL: NCT06976606
Title: An Observational Study to Assess Real-world Patient Characteristics, Clinical Course, and Treatment Patterns for Symptomatic Patients With Arrhythmogenic Cardiomyopathy (ACM) Due To a PlaKoPhilin-2 Pathogenic Variant (PKP2)
Brief Title: A Study to Assess Real-world Patient Characteristics and Clinical Course for Symptomatic Patients With PKP2-ACM
Acronym: SNAPSHOT- PKP2
Status: Recruiting | Type: Observational
Sponsor: Lexeo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: LX2020-03
Record Dates: First submitted 2024-03-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Arrhythmogenic Cardiomyopathy; PKP2-ACM; PKP2-ARVC
Keywords: Arrhythmogenic Cardiomyopathy; ACM; Cardiomyopathy; ARVC; Arrhythmogenic Right Ventricular; Arrhythmogenic Right Ventricular Dysplasia; Genetic cardiomyopathy; Gene Therapy; PKP2 Gene; Plakophilin-2; LX2020; SNAPSHOT-PKP2; Ventricular Arrhythmia; PVCs; Sudden Cardiac Death; Cardiac Arrest
MeSH Terms: conditions — Cardiomyopathies; Arrhythmogenic Right Ventricular Dysplasia; Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples will be collected to assess cardiac biomarkers associated with PKP2-ACM and to study existing antibodies to AAVrh.10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
An observational study to assess real-world patient characteristics and clinical course of disease in participants with PKP2-ACM.

DETAILED DESCRIPTION:
SNAPSHOT-PKP2 is an observational, multicenter study that consists of 2 parts, a retrospective EMR review (up to 2 years) and a prospective observational study (1 year), to evaluate the clinical burden of illness of patients with PKP2-ACM, and to prospectively evaluate changes in key cardiac parameters and patient-reported outcome measures (PROMs) associated with PKP2-ACM progression.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a clinical diagnosis of ACM as defined by the 2010 revised Task Force Criteria (TFC)
* Documentation of a pathogenic or likely pathogenic truncating variant in PKP2
* Frequent premature ventricular contractions (PVCs)
* Patients must have an ICD placed prior to enrollment
* Left ventricular ejection fraction (LVEF) ≥ 50% for Part A participants. Left ventricular ejection fraction (LVEF) ≥40% for Part B participants.

Exclusion Criteria:

* Evidence of variant(s) in addition to PKP2 that meet standard criteria to be considered pathogenic or likely pathogenic for an arrhythmogenic cardiomyopathy.
* A history of other cardiac abnormalities as specified in the protocol.
* New York Heart Association symptoms of heart failure of Class IV at the time of consent.
* A history of prior gene transfer therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years at time of consent with confirmed diagnosis of ACM and documentation of PKP2 variant.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Premature ventricular contractions (PVC) | 12 months
  Change from baseline

SECONDARY OUTCOMES:
Ventricular arrhythmias and associated clinical events | 12 months
  Change from baseline by interrogation of implanted cardioverter defibrillator and remote cardiac monitoring
ECG parameters | 12 months
  Change from baseline
Cardiac structure and function | 12 months
  Change from baseline via cardiac MRI and echocardiogram
Patient reported outcomes | 12 months
  Patients' Global Impression of Change (PGIC) scale, measuring participant perception of change from baseline.
Patient reported outcomes | 12 months
  Patients' Global Impression of Severity (PGIS) scale, measuring patient perception of disease progression.
Cardiac Biomarkers | 12 months
  Change from baseline
Health resource utilization | 12 months
  Number of ED, urgent care and outpatient visits, and hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Lexeo Clinical Trials, Study Director — Lexeo Therapeutics
Locations (6):
- United States (6):
  - Leland Stanford Junior University, Redwood City, California
  - Johns Hopkins University, Baltimore, Maryland
  - Northshore University Healthsystem Research Institute, Columbia, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No